CLINICAL TRIAL: NCT06357585
Title: Evaluation of the Effect of Web-Based Education Provided to Parents of Children With Leukemia on Parents' Knowledge Level, Satisfaction and Self-Efficacy
Brief Title: Providing Web-based Training to Parents Of Children With Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBUBURCUCALİK
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-04

CONDITIONS: Leukemia
Keywords: leukemia; child; nurses
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Intervention Model Description: Web-based training will be provided to parents in the experimental group, and parents in the control group will continue their routine treatment and care process.
Who Masked: Participant
Masking Description: Participant blinding was done because the parents who participated in the study voluntarily did not know which group they were in until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web based education group (Experimental): Parents in the experimental group will be given web-based training for 5 weeks.
  Interventions: Other: Web based education
- control group (Experimental): No intervention will be made to the parents in the control group, and the children will continue their routine care and treatment process.
  Interventions: Other: inactive group

INTERVENTIONS:
Other: Web based education — Web-based training will be provided to the parents in the experimental group regarding care practices for children diagnosed with leukemia.
  Arms: web based education group
Other: inactive group — Parents in the control group will continue to receive routine care and treatment.
  Arms: control group

SUMMARY:
Following and implementing innovations and current developments in care practices for children diagnosed with leukemia and their parents will allow the quality of care to increase. The purpose of this research is to evaluate the effect of web-based education given to parents of children diagnosed with leukemia on their knowledge level, satisfaction and self-efficacy.

The research is a single-blind randomized controlled experimental research type. The research will be conducted in a single center, Ankara Bilkent City Hospital MH4 Children's Hospital Hematology-Oncology Clinics and Leukemia Polyclinic. The population of the research consists of parents of children diagnosed with leukemia between the ages of 2-18 who are followed and treated in the specified places. The sample of the research consists of 72 participants, 36 in the experimental group (the group that received web-supported training) and 36 in the control group (the group that continued routine treatment).

The consent of the parents who meet the research criteria and voluntarily agree to participate in the study will be obtained with the "Informed Voluntary Consent Form" and the parents in both the experimental group and the control group will be given the "Child and Parent Introductory Information Form", "Child with Leukemia Parent Information Level Pre-Test Evaluation Form". ", "Generalized Perceived Self-Efficacy Scale" will be applied. Once the sufficient number is reached, web-based training will be provided to the parents in the experimental group. "Parents of Children with Leukemia Knowledge Level Post-Test Evaluation Form", "Generalized Perceived Self-Efficacy Scale" and "Web-Based Parents of Children with Leukemia Training Satisfaction Evaluation Form" will be applied to the parents who complete the training. No intervention will be made to the parents in the control group, and the children will continue their routine care and treatment process. The "Child with Leukemia Parent Knowledge Level Posttest Evaluation Form" and the "Generalized Perceived Self-Efficacy Scale" will also be applied to the parents in the control group.

DETAILED DESCRIPTION:
Leukemia is one of the most common types of cancer among pediatric cancers. A diagnosis of leukemia affects both children, parents and all individuals who interact with the child, and can cause physical, social, spiritual and economic problems.

In childhood cancers, parent education is one of the important nursing practices that must be carried out so that parents can feel competent in care practices and the child can be given the most appropriate care in line with their needs. The content of these trainings should focus on parents gaining skills by participating in care. It is important to provide quality education to parents with methods that suit their learning preferences and styles. As the use of technology has gained importance around the world, technology-based interventions for children and parents have also become important. Developments in the field of digital health can make it easier to transfer many aspects of cancer treatment into families' lifestyles with new options. Technology-based interventions contribute to children and parents as they provide opportunities such as appealing to different senses and providing continuous access to information. One of these interventions is the creation of web-based programs. Carrying out training via web bases provides the opportunity to easily access training content without any time or space limitation. It also allows the individual to determine his own learning pace and examine the materials easily.

Patients and their relatives often use the internet to access cancer-related information. However, some of the information on the internet, which is an easy and fast way to access information, may be outdated or inaccurate. Although the use of the internet as an alternative method of accessing information and the fact that it is a fast and easy method of accessing information is seen as a great advantage in terms of health services, inaccurate and outdated information on the website poses a major problem. Therefore, it is important to create websites where parents can access accurate and up-to-date information.Following and implementing innovations and current developments in care practices for children diagnosed with leukemia and their parents will allow to increase the quality of care. The purpose of this research is to evaluate the effect of web-based education given to parents of children diagnosed with leukemia on their knowledge level, satisfaction and self-efficacy.

The hypotheses of the research are presented below; HOa: There is no difference between the knowledge levels of parents who received web-based child care training with a diagnosis of leukemia and the knowledge levels of parents who did not receive training.

HOb: There is no difference between the self-efficacy scale scores of parents who received web-based leukemia child care training and the self-efficacy scale scores of parents who did not receive training.

H1a: There is a difference between the knowledge levels of parents who received web-based child care training with a diagnosis of leukemia and the knowledge levels of parents who did not receive training.

H1b: There is a difference between the self-efficacy scale scores of parents who received web-based leukemia child care training and the self-efficacy scale scores of parents who did not receive training.

The research is a single-blind randomized controlled experimental research type, and "pretest-posttest randomized control group design", one of the experimental research types, will be used in the research. The research will be conducted in a single center, Ankara Bilkent City Hospital MH4 Children's Hospital Hematology-Oncology Clinics and Leukemia Polyclinic. The population of the research consists of parents of children diagnosed with leukemia between the ages of 2-18 who are followed and treated in the specified places. "Simple random sampling method" will be used in sample selection. Before starting the research, the sample size was determined with the Power and Sample size analysis G Power Program. Medium effect size f = 0.25, Type I error: 0.05, Type II error: 80% (power), and the number of samples calculated was 17 parents for the group receiving web-supported education (experimental group), 17 parents for the group receiving routine care. For the group (control group), 17 parents were determined as a total of 34 parents. However, it was planned to conduct the research with a total of 60 parents, 30 parents for both groups, in order to avoid problems in population generalization, to fulfill the parametric test assumptions of the research, and to reveal the relationships between variables more clearly. Considering that there may be losses due to the research requiring long-term follow-up, 72 parents will be included in the research by taking 20% more than the determined sample number. In the randomization to be carried out, the "simple randomization method" will be used in order to provide equal samples for both groups (experiment-control).

In order to collect data in the research, "Child and Parent Introductory Information Form", "Child with Leukemia Parent Information Level Pre-Test-Post-Test Evaluation Form", "Web-Based Child with Leukemia Parent Education Satisfaction Evaluation Form", "Generalized Perceived Self-Efficacy Scale" will be used. The consent of the parents who meet the research criteria and voluntarily agree to participate in the study will be obtained with the "Informed Voluntary Consent Form" and the parents in both the experimental group and the control group will be given the "Child and Parent Introductory Information Form", "Child with Leukemia Parent Information Level Pre-Test Evaluation Form". ", "Generalized Perceived Self-Efficacy Scale" will be applied. Parents who meet the research criteria and voluntarily agree to participate in the study will be included in the experimental and/or control group according to the randomization list. Once the sufficient number is reached, the parents in the experimental group will be contacted via mobile phone and necessary explanations (name of the site, membership to the site, how to log in to the site, menus on the site and how to use these menus, link of the site, training duration) will be made. In order for users to learn according to their own learning levels, without space and time constraints, 5 modules prepared in line with the objectives and achievements, 5 video lectures related to the modules, and videos showing the applications in the video lectures will be uploaded to the site. Before the modules are uploaded to the website, expert opinion will be obtained and necessary arrangements will be made. Training achievements and objectives will be given in the introduction part of the modules, and brief information on the subject will be given at the beginning of the video.

Users will be asked to review the relevant modules and videos, and after reviewing the modules, they will be asked to tick the "I have read and understood" box. Parents in the experimental group will be given web-based training for 5 weeks. "Parents of Children with Leukemia Knowledge Level Post-Test Evaluation Form", "Generalized Perceived Self-Efficacy Scale" and "Web-Based Parents of Children with Leukemia Training Satisfaction Evaluation Form" will be applied to the parents who complete the training. No intervention will be made to the parents in the control group, and the children will continue their routine care and treatment process. At the end of 5 weeks, "Child with Leukemia Parent Knowledge Level Posttest Evaluation Form" and "Generalized Perceived Self-Efficacy Scale" will also be applied to the parents in the control group. At the end of the study, the modules will be shared with the control group.

To conduct the research, the necessary written permissions were obtained from the Ankara Provincial Health Directorate with the permission of the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being 18 years or older,
* Being directly responsible for the child's care,
* Not having any physical or mental illness,
* Being able to use a computer or mobile phone,
* Having internet access and being able to use the internet,
* Being open to communication,
* Being literate,
* Being able to speak and understand Turkish.

Exclusion Criteria:

* Not following the site of membership,
* Not having internet access and not being able to use the internet,
* Being a foreign national,
* Having vision or hearing problems,
* Being illiterate,
* To give up participating in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Child with Leukemia Parent Knowledge Level Pre-Test Evaluation Form | at the time before pre-education
  This form aims to evaluate the parents' knowledge levels before the training and the effectiveness of the training given in the post-training period. The form consists of "19" closed-ended questions about common symptoms in children with leukemia and the management of these symptoms. The evaluation form before the training (pre-test) and after the training (post-test) consists of the same questions. All of the items in questions 1, 2, 3, 6, 7, 8, 9, 11, 13, 14, 15, 16, 17, 18, 19 are correct, and questions 4, 5, 10 and 10 are correct. There is only one correct answer to question 12. Each of the items in questions 1, 2, 3, 6, 7, 8, 9, 11, 13, 14, 15, 16, 17, 18, 19 is worth 1 point, and "water and soap" in question 4 is worth 1 point. 5 points. The total knowledge score for the correct answers to the questions "once a week", 25,000 mm3 in the 10th question and "4-6 times" in the 12th question will be calculated as 1 point each.
Child with Leukemia Parent Knowledge Level Post-Test Evaluation Form | within 15 days after education
  This form aims to evaluate the parents' knowledge levels before the training and the effectiveness of the training given in the post-training period. The form consists of "19" closed-ended questions about common symptoms in children with leukemia and the management of these symptoms. The evaluation form before the training (pre-test) and after the training (post-test) consists of the same questions. All of the items in questions 1, 2, 3, 6, 7, 8, 9, 11, 13, 14, 15, 16, 17, 18, 19 are correct, and questions 4, 5, 10 and 10 are correct. There is only one correct answer to question 12. Each of the items in questions 1, 2, 3, 6, 7, 8, 9, 11, 13, 14, 15, 16, 17, 18, 19 is worth 1 point, and "water and soap" in question 4 is worth 1 point. 5 points. The total knowledge score for the correct answers to the questions "once a week", 25,000 mm3 in the 10th question and "4-6 times" in the 12th question will be calculated as 1 point each.
Web-Based Child with Leukemia Parent Education Satisfaction Evaluation Form | within 15 days after education
  This form has been prepared to determine the objectives for the experimental class, the website provided for the training of the participants, and the training contents. There are "43" statements in the form, which include evaluation of the appearance of the website, its usability, the content of the website and the training provided on the website, and the level of usefulness. "18" expression in the form is prepared for the appearance and usability of the website, "12" expression is for the video explanations on the website, and "13" expression is for the modules on the website. The form was prepared according to the five-point Likert type (1 = Strongly Disagree, 2 = Disagree, 3 = Neither Agree nor Disagree, 4 = Agree, 5 = Strongly Agree). The lowest score from the form is "43" and the highest score is "215". A high score is considered to indicate that parents are satisfied with the education provided.
Generalized Perceived Self-Efficacy Scale | at the time before pre-education
  This scale aims to determine the amount of self-efficacy level of web-supported education given to children with leukemia. Scale items receive scores between 1 and 4, consist of positive items, and are evaluated based on the total score. Grading of the scale; Not true (1), somewhat true (2), more true (3), completely true (4). Total score is between 10-40. High score is considered as high self-efficacy perception.
Generalized Perceived Self-Efficacy Scale | at the within 15 days after education
  This scale aims to determine the amount of self-efficacy level of web-supported education given to children with leukemia. Scale items receive scores between 1 and 4, consist of positive items, and are evaluated based on the total score. Grading of the scale; Not true (1), somewhat true (2), more true (3), completely true (4). Total score is between 10-40. High score is considered as high self-efficacy perception.

CONTACTS AND LOCATIONS:
Overall Officials: BURCU ÇALIK BAĞRIYANIK, Principal Investigator — University of Health science
Locations (1):
- University of Health Sciences, Ankara, Keçiören, Turkey (Türkiye)